CLINICAL TRIAL: NCT07304245
Title: The Asymmetry of Endometriotic Lesions as Demonstration of the Theory of Menstrual Reflux and Anatomical Niches: Italian Multicenter Study by the ETIC Group
Brief Title: The Asymmetry Distribution of Endometriotic Lesions: Italian Multicenter Study
Acronym: NICCHIENDO
Status: Completed | Type: Observational
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 0029787 U; NICCHIENDO (Other: IRCCS Fondazione Ca' Granda, Ospedale Maggiore, Policlinico, Milan)
Record Dates: First submitted 2024-08-19; First posted 2025-12-26 (Actual); Last update posted 2025-12-26 (Actual); Status verified 2025-10

CONDITIONS: Analyze the Laterality of Endometriotic Lesions and Endometriosis-related Tumors; Endometriosis
MeSH Terms: conditions — Endometriosis | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: surgery — All patients enrolled in the study underwent surgery for endometriosis between 2013 and 2023.

SUMMARY:
This study aims to understand whether endometriosis lesions - and tumors that can arise in association with endometriosis - occur more often on one side of the pelvis than the other.

During surgery, doctors will record the exact location of each lesion to see if there is a consistent right- or left-sided pattern.

Understanding these patterns may help improve knowledge about how endometriosis develops (pathogenesis), and thus improve its treatment.

ELIGIBILITY:
Inclusion Criteria:

* age ≥18 years at the time of histological diagnosis of endometriosis
* patients undergoing surgery with endometriotic lesions or patients with endometriotic lesions associated with endometrioid or clear cell ovarian cancer (Stage I-II) or borderline seromucinous ovarian cancer
* first operation for endometriosis in the reference center (if recurrence consider only if both operations were performed at the reference center).

Exclusion Criteria:

* age <18 years
* patients affected by Stage I-II endometrioid or clear cell carcinoma or seromucinous borderline ovarian cancer not associated with endometriosis or in a more advanced stage of disease
* women with an ultrasound diagnosis of endometriosis who have not undergone surgery
* previous operations for endometriosis performed at another center

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients with histological diagnosis of endometriosis and endometriosis associated with endometrioid carcinoma, clear cell carcinoma and seromucinous borderline tumor operated at the Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico and at the centers participating in the study from 01/2013 to 12/2023 will be recruited.
  Data relating to histological diagnosis will be collected from medical records.
  In particular, in addition to tumours associated with endometriosis, data will be collected from patients with a histological diagnosis of:
  1. ovarian endometriosis
  2. intestinal endometriosis
  3. ureteral endometriosis
  4. sciatic nerve endometriosis
  5. inguinal-round ligament endometriosis
  6. uterosacral ligament endometriosis
  7. peritoneal endometriosis
  8. diaphragmatic endometriosis
  9. pleural and pulmonary endometriosis
  10. umbilical endometriosis (associated with right hemidiaphragm and/or left hemidiaphragm)
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Actual)
Dates: Start 2024-09-01 (Actual); Primary Completion 2025-05-01 (Actual); Study Completion 2025-07-01 (Actual)

PRIMARY OUTCOMES:
Asymmetric distribution of endometriotic lesions on paired pelvic organs | At the time of index surgery
  Proportion of patients presenting an asymmetric (right- or left-sided) distribution of endometriotic lesions on even and symmetrical pelvic organs (e.g., ovaries, uterosacral ligaments), based on the laterality observed and described during the index surgical procedure.
  Side-specific frequencies (right vs left) will be reported as number and percentage.

SECONDARY OUTCOMES:
Asymmetric distribution of malignant ovarian lesions related to endometriosis | At the time of index surgery
  Proportion of patients presenting an asymmetric (right- or left-sided) distribution of malignant lesions related to endometriosis-specifically endometrioid ovarian carcinoma, clear cell ovarian carcinoma, and seromucinous borderline tumors-based on the laterality observed and described during the index surgical procedure.
  Side-specific frequencies (right vs left) will be reported as number and percentage.

CONTACTS AND LOCATIONS:
Locations (1):
- Gynecology Unit, IRCCS Fondazione Ca' Granda Ospedale Maggiore Policlinico, Milan, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided